CLINICAL TRIAL: NCT06936943
Title: A Multicenter, Open-label, Uncontrolled Study to Evaluate the Efficacy and Safety of ONO-4538 in Patients With Richter's Transformation
Brief Title: ONO-4538 Study in Patients With Richter's Transformation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4538-131; jRCT2071250005 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Richter's Transformation
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ONO-4538 (Experimental): ONO-4538 480 mg solution administered intravenously every 4 weeks
  Interventions: Drug: ONO-4538

INTERVENTIONS:
Drug: ONO-4538 — every 4 weeks
  Other Names: Nivolumab; Opdivo

SUMMARY:
Investigate the efficacy and safety of ONO-4538 in patients with Richter's transformation

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of diffuse large B-cell lymphoma (DLBCL)-type or Hodgkin lymphoma(HL)-type Richter's transformation with a history of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL)
* In the case of DLBCL-type Richter's transformation, refractory, intolerant or ineligible for treatment of DLBCL
* Patients with measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Expected to survive for 90 days or more

Exclusion Criteria:

* Serious complications
* Active multiple cancers
* Active central nervous system (CNS) disease
* History of allogeneic hematopoietic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) (Centralized assessment) | up to 4 years

SECONDARY OUTCOMES:
Objective response rate (ORR) (site investigator assessment) | up to 4 years
Overall survival (OS) | up to 4 years
Progression free survival (PFS) | up to 4 years
Disease control rate (DCR) | up to 4 years
Duration of response (DOR) | up to 4 years
Time to response (TTR) | up to 4 years
Best overall response (BOR) | up to 4 years
Change rate from baseline in the sum of diameters (SPD) of target lesions | up to 4 years
Best change rate from baseline in the sum of diameters (SPD) of target lesions | up to 4 years
Improvement rate of B symptom | up to 4 years
Safety (Adverse event) | Up to 30 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (9):
- Japan (9):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Kyusyu University Hospital, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kyoto University Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō-Ku, Tokyo
  - National Cancer Center Hospital, Chuo Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No